CLINICAL TRIAL: NCT06149208
Title: PROSPR: PeriopeRative Opioid Stewardship Program of Research (Phase 5 - ED Discharge Study)
Brief Title: Emergency Department Discharge for Type II Supracondylar Fractures - PROSPR Phase 5
Status: Not yet recruiting | Type: Observational
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Conor McDonnell, Principal Investigator, Associate Professor, The Hospital for Sick Children
Other Study IDs: 1000080963
Record Dates: First submitted 2023-11-20; First posted 2023-11-28 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: Supracondylar Fracture
MeSH Terms: interventions — Interviews as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Year 1 - Treatment Change: This group will receive the new treatment standard
  Interventions: Behavioral: Interview
- Year 2 - Sustainability: This group will be used to measure sustainability of the new treatment standard
  Interventions: Behavioral: Interview

INTERVENTIONS:
Behavioral: Interview — Families will complete interviews about their experiences with the new treatment standard and managing pain at home

SUMMARY:
The knowledge that patients will not suffer untreated pain at home is central to managing supracondylar fracture (SCF) patients on an outpatient basis at a time of limited healthcare resources. The investigators hypothesize that children with uncomplicated Type II supracondylar fractures (SCF) can be sent home from the Emergency Department (ED) in a temporary cast, and that fracture pain can be safely managed opioid-free at home both before and after surgical repair. The investigators further hypothesize that managing such patients on an ambulatory out-patient basis will increase hospital-bed availability without compromising surgical outcomes.

DETAILED DESCRIPTION:
Since January 2020, some 1050 admission-days have been accountable to Type II SCF with a mean stay of 1.2 days (SD 0.52) in this institution. However, some patients spend more than 48-hours in-house awaiting surgery, often with two periods of fasting greater than 8-hours imposed, due to competing interests with higher priority cases on the OR's shared add-on board. These patients occupy a hospital bed at a time when resources are severely depleted. The COVID pandemic has enforced many stressors on healthcare across Ontario and one mitigation for same was the diversion of pediatric admissions from surrounding community hospitals to HSC to create 'extra beds' for acute adult admissions in the community. This diversion has imposed significant bed-demands on HSC and with COVID-related admission rates in the community decreasing it has proved difficult to re-route routine pediatric admissions (such as SCF) to the community. This institution's Pediatric Intensive Care Unit (PICU) has been operating above capacity for some time now leading to 'controlled slowdowns' in elective operative procedures, resulting in months of cancellation of some 40-75% of elective pediatric surgery.

This institution's PROSPR program delivered standardization of opioid prescribing at hospital discharge post pediatric SCF repair. Since 2021 the investigators decreased overprescribing of opioids to SCF patients at hospital discharge to the tune of 360%. This work has also created pathways for safe return and disposal which decreased MME amount of opioid lost to follow-up in the community by over 500%. The investigators also demonstrated that home consumption of morphine is so low that it is feasible to completely remove opioid prescribing from pediatric SCF discharge planning which opens the possibility of managing surgical scheduling on an out-patient basis whererby families will derive increased satisfaction from being able to wait at home for surgery.

ELIGIBILITY:
Inclusion Criteria:

* requiring surgery for Type II supracondylar fracture

Exclusion Criteria:

* none

Max Age: 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: All children meeting eligibility criteria at our institution over the next two years (2023-2025) will be approached for consent
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-28 (Estimated)

PRIMARY OUTCOMES:
Decreasing opioid prescribing to zero 0 - year 1 | From ED Discharge through to post-operative discharge (approximately 1 week)
  Patient prescriptions will be reviewed to ensure no opioids were erroneously prescribed
Decreasing opioid prescribing to zero 0 - year 2 | From ED Discharge through to post-operative discharge (approximately 1 week)
  Patient prescriptions will be reviewed to ensure no opioids were erroneously prescribed

SECONDARY OUTCOMES:
Reduced hospital bed occupancy - year 1 | End of Year 1
  Bed allocation rates will be compared to those obtained prior to the study commencing
Reduced hospital bed occupancy - year 2 | End of Year 2
  Bed allocation rates will be compared to those obtained prior to the study commencing and compared to year 1
Improved family experience after discharge from Emergency Department (ED) - year 1 | 2 Days post-ED discharge - year 1
  Families will complete a semi-structured interview detailing their experience with managing the child's pain at home since ED discharge
Improved family experience after discharge post-operatively - year 1 | 3-5 Days post-operative discharge - year 1
  Families will complete a semi-structured interview detailing their experience with managing the child's pain at home since post-operative discharge
Improved family experience after discharge from Emergency Department (ED) - year 2 | 2 Days post-ED discharge - year 2
  Families will complete a semi-structured interview detailing their experience with managing the child's pain at home since ED discharge
Improved family experience after discharge post-operatively - year 2 | 3-5 Days post-operative discharge - year 2
  Families will complete a semi-structured interview detailing their experience with managing the child's pain at home since post-operative discharge
Reduced need for follow-up xrays - year 1 | 3 Weeks post-operative discharge - year 1
  The number of follow-up xrays required at clinic check-in will be compared to the average number of x-rays required at clinic check-in prior to the commencement of the study
Reduced need for follow-up xrays - year 2 | 3 Weeks post-operative discharge - year 2
  The number of follow-up xrays required at clinic check-in will be compared to the average number of x-rays required at clinic check-in prior to the commencement of the study and to year 1

CONTACTS AND LOCATIONS:
Overall Officials: Conor Mc Donnell, Principal Investigator — Staff Anesthesiologist
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No